CLINICAL TRIAL: NCT01266213
Title: Randomized Phase II Study OF Goserelin (G) Plus Fulvestrant (F) vs. G Plus Anastrozole (A)vs. G Alone for HR+, Tamoxifen Pretreated, Premenopausal Woman
Brief Title: Fulvestrant (F)/Goserelin (G) vs Anastrozole (A)/G vs G for Premenopausal Women
Acronym: FLAG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Asan Medical Center (Other); Seoul National University Hospital (Other); Severance Hospital (Other); Ulsan University Hospital (Other); Kosin University Gospel Hospital (Other); Korea University Guro Hospital (Other); Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Young-Hyuck Im, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-04-001
Record Dates: First submitted 2010-12-19; First posted 2010-12-24 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Breast Cancer; Estrogen Receptor Positive Tumor; Breast Cancer Nos Premenopausal
Keywords: fulvestrant; anastrozole; goserelin; tamoxifen; premenopausal; hormone receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Goserelin; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fulvestrant plus Goserelin (Experimental)
  Interventions: Drug: Fulvestrant plus Goserelin; Drug: Anastrozole plus Goserelin; Drug: Goserelin
- Anastrozole plus Goserelin (Experimental)
  Interventions: Drug: Fulvestrant plus Goserelin; Drug: Anastrozole plus Goserelin; Drug: Goserelin
- Goserelin alone (Active Comparator)
  Interventions: Drug: Fulvestrant plus Goserelin; Drug: Anastrozole plus Goserelin; Drug: Goserelin

INTERVENTIONS:
Drug: Fulvestrant plus Goserelin — Fulvestrant s.c. plus Goserelin s.c.
  Other Names: Anastrozole plus Goserelin
Drug: Anastrozole plus Goserelin — Anastrozole 1 mg p.o. plus Goserelin s.c.
  Other Names: Fulvestrant plus Goserelin
Drug: Goserelin — Goserelin s.c.
  Other Names: Fulvestrant plus Goserelin; Anastrozole plus Goserelin

SUMMARY:
Fulvestrant is an ER antagonist with no agonist effects, which binds, blocks and degrades the ER. Fulvestrant is comparable to third-generation aromatase inhibitors in terms of efficacy and tolerability for patients who have progressed on prior tamoxifen therapy and past studies have found all three-third-generation AIs to be at least as good as tamoxifen in first-line metastatic therapy in postmenopausal women. Fulvestrant has been studied little in premenopausal women despite of its attractive mechanism of actions. The clinical effectiveness of fulvestrant as a treatment for advanced breast cancer has previously been demonstrated at the standard dose (AD; 250 mg/mo) in several phase III clinical trials in postmenopausal women. However, there is evidence to suggest that doses of fulvestrant higher than 250 mg may have greater pharmacodynamic activity against the ER pathway. Moreover, dose-dependent clinical activity has been observed for fulvestrant. The activity of a fulvestrant high-dose (HD; 500 mg/mo) regimen has been investigated in two recent studies. A pilot Japanese study showed fulvestrant HD to have clinical activity in the treatment of advanced or recurrent breast cancer, to be well tolerated, and to result in plasma levels approximately double those seen with fulvestrant low-dose. Subsequently, a neoadjuvant study comparing fulvestrant low-dose and high-dose reported that significantly greater Ki67 and ER downregulation was achieved with the high-dose compared with the low-dose regimen and that both doses were well tolerated. A recent randomized trial also showed superior outcome of high-dose fulvestrant than AI.

Based on this rationale, we introduced high-dose fulvestrant with LHRH agonist as a randomized trial comparing with AI plus LHRH agonist and LHRH alone in premenopausal metastatic breast cancer patients who failed to tamoxifen treatment.

DETAILED DESCRIPTION:
This randomized phase II trial is studying fulvestrant with goserelin for ovarian suppression by goserelin to see how well it works compared to anastrozole with goserelin and goserelin alone in recurrent or metastatic ER-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1) All patients must be female and premenopausal. Premenopausal is defined as either: ① last menstrual period within 3 months, or ② post-hysterectomy without bilateral oophorectomy and with FSH in the premenopausal range (≤ 30 mIU/mL), or, ③ if on tamoxifen within the past 3 months, a plasma estradiol in the premenopausal range (≥20 pg/mL), ④ if in case of chemotherapy induced amenorrhea, a plasma estradiol in the premenopausal range (≥20 pg/mL).

  2) Patients must have either positive estrogen and/or progesterone receptor determination by IHC or competitive binding assay on metastatic disease, or if not performed on their metastatic disease a positive result on their primary breast cancer specimen.

  3) No HER2 overexpressing breast cancer by IHC 3+ or FISH. 4) Patients who showed progressive disease on tamoxifen treatment as a palliative hormonal therapy or an adjuvant endocrine treatment 5) Patients who recurred after 5 years of tamoxifen use and could not be considered for resume to tamoxifen treatment.

  6) No prior treatment with an aromatase inhibitor or inactivator or fulvestrant 7) No prior treatment with an LH/RH agonist/antagonist except the use for ovarian protection for 6 months during adjuvant chemotherapy.

  8) No adjuvant chemotherapy within 1 year of study entry. 9) Patients must have an ECOG performance status of 0, 1, or 2. 10) Patients must have adequate bone marrow, hepatic, and renal function 11) Patients must not have received chemotherapy or hormonal therapy for at least 4 weeks prior to enrollment.

  12) Patients may receive irradiation to any bony sites of disease for pain control or for prevention of fracture.

  13) Patients may continue on bisphosphonates who already established on bisphosphonate therapy for at least 3 months.

  14) Patients who are pregnant or lactating are ineligible. Must be using effective contraception or not be of childbearing potential.

  15) Patients must not have had an active malignancy other than breast cancer, in situ carcinoma of the cervix, or non-melanomatous skin cancers in the past 5 years.

  16) No active, unresolved infection. 17) All patients must give signed written informed consent

Exclusion Criteria:

1. Patients who had received previous treatment for metastatic disease (including systemic cytostatic or hormonal treatment) other than tamoxifen.
2. Lymphangitic pulmonary metastases
3. Multiple or diffuse hepatic metastases
4. Documented parenchymal or leptomeningeal brain metastasis
5. HER-2 overexpressing breast cancer and concomitant trastuzumab treatment is not allowed
6. Serious uncontrolled intercurrent infections
7. Serious intercurrent medical or psychiatric illness, including active cardiac disease
8. Pregnancy or breast feeding
9. Second primary malignancy (except in situ carcinoma of the cervix or resected papillary thyroid carcinoma or adequately treated nonmelanomatous carcinoma of the skin or other malignancy treated at least 5 years previously with no evidence of recurrence)

Max Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 147 (Estimated)
Dates: Start 2010-12; Primary Completion 2018-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Time to Progression (TTP) | from the date of therapy to the date of progression every 3 months
  To measure TTP, disease status will be measured every 3 cycles or clinically documented till progression

SECONDARY OUTCOMES:
overall response | after 3 months from the first date of therapy
  Before start of 4th cycle of therapy, outcome measure will be perfomred to evaluate response
overall survival | from the first date of therapy till death
  from time to the first day of therapy to death
Toxicity | from the first date of therapy to death every cycle of therapy (monthly)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hyuck Im, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim JY, Im SA, Jung KH, Ro J, Sohn J, Kim JH, Park YH, Kim TY, Kim SB, Lee KS, Kim GM, Kim SH, Kim S, Ahn JS, Lee KH, Ahn JH, Park IH, Im YH; breast cancer committee of Korean Cancer Study Group (KCSG). Fulvestrant plus goserelin versus anastrozole plus goserelin versus goserelin alone for hormone receptor-positive, HER2-negative tamoxifen-pretreated premenopausal women with recurrent or metastatic breast cancer (KCSG BR10-04): a multicentre, open-label, three-arm, randomised phase II trial (FLAG study). Eur J Cancer. 2018 Nov;103:127-136. doi: 10.1016/j.ejca.2018.08.004. Epub 2018 Sep 14. PMID 30223226
- See also: Korea Cancer Study Group — http://kcsg.org